CLINICAL TRIAL: NCT01283737
Title: A Randomized, Subject-blind, Controlled Pilot Trial to Evaluate the Effectiveness and Safety of the Use of Demineralized Bone Matrix (DBX®) Versus Mosaicplasty in the Treatment of Late-Stage Osteochondritis Dissecans (OCD) of the Knee in Patients With a Mature Skeleton
Brief Title: Use of Demineralised Bone Matrix (DBX) in Osteochondritis Dissecans (OCD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Synthes GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-BIO-T-XX-001-01
Record Dates: First submitted 2010-05-28; First posted 2011-01-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Osteochondritis Dissecans
Keywords: Osteochondritis Dissecans; OCD; Mosaicplasty; Demineralised Bone Matrix; DBX; DBX Putty
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBX (Experimental): DBX Putty in glass syringe
  Interventions: Device: DBX Putty
- Mosaicplasty (Active Comparator)
  Interventions: Procedure: Mosaicplasty

INTERVENTIONS:
Device: DBX Putty — OCD of the knee will be treated with DBX Putty
  Arms: DBX
Procedure: Mosaicplasty — Mosaicplasty procedure performed to treat OCD of the knee
  Arms: Mosaicplasty

SUMMARY:
This is a 1:1 randomised pilot study in 30 patients in 1 site in Helsinki, Finland.

The investigators hypothesize that function, pain, type and quality of cartilage in adult patients with osteochondritis dissecans of the knee will be better in the DBX group compared to the mosaicplasty group.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age between 18 years and 65 years
* Females of childbearing potential must have a negative serum or urine pregnancy test at the time of inclusion
* Females of childbearing potential must be willing to use effective means of birth control for at least 1 year post surgery. Medically acceptable contraceptives include:

  1. Surgical sterilisation
  2. Approved hormonal contraceptives
  3. Barriers methods combined with a spermicide
  4. An intrauterine device
  5. Abstinence alone is not considered an acceptable method of contraception
* Late stage Osteochondritis Dissecans (ICD-10 code M93.2) of the knee classified as stage III or IV (Anderson MRI classification)
* Mature skeleton
* Written informed consent prior to any study specific procedures (except the procedures necessary to determine eligibility)
* Ability and willingness to comply with all study specific procedures, including attending all follow-up visits up to 12 months postoperative and completing questionnaires in a local language

Exclusion Criteria:

* More than 1 knee affected
* Patients who can be treated with conservative treatment alone, unless there is evidence of at least 6 months failed previous treatment
* Systemic disease including AIDS, HIV, Hepatitis or any other disease that would prevent normal organ and marrow function.
* Patients undergoing systemic cortisone treatment or immunosuppressive therapy (e.g. avascular necrosis)
* Patients undergoing active cancer therapy (chemotherapy, radiation treatment).
* History of alcohol abuse or illegal drug use.
* Participation in any other device or drug trial within 3 months prior to the inclusion in the study
* Presence of at least one contraindication for DBX® Putty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change of Brittberg-Peterson functional assessment score from baseline until 12 months post-op | At enrollment (day -7), at full weight-bearing (6-8 weeks post-operative), 6 months post-operative, 12 months post-operative
  Score 0-130 (see Clin Orthop Relat Res 2000 May;374:212-34) to assess function and pain

SECONDARY OUTCOMES:
Type and quality of the formed cartilage to assess the effectiveness of the treatment | 12 months post-operative
  The type and quality of the newly formed cartilage will be assessed with arthroscopy and/or MRI /dGEMRIC)
Number of patients with complications to assess the safety of the use of the treatment | Enrolment (day -7) until 12 months post-operative
  All adverse events and complications will be recorded throughout the trial and assessed for severity and causality.

CONTACTS AND LOCATIONS:
Overall Officials: Jari Salo, MD, Principal Investigator — Töölö Hospital
Locations (1):
- Töölö Hospital, Helsinki, Finland